CLINICAL TRIAL: NCT02316301
Title: Optimal Timing of Misoprostol Administration Prior to Office Hysteroscopy; a Randomized Controlled Trial.
Brief Title: Optimal Timing of Misoprostol Administration Prior to Office Hysteroscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Usama M Fouda, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Long miso/short miso/hyst
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Pain
Keywords: Misoprostol, pain, office hysteroscopy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Long interval misoprostol (Experimental): A small envelope including two labeled plastic bags (A & B) (each bag containing either 2 misoprostol tablets(400µg) or 2 identically appearing placebo tablets) will be packaged in sequentially numbered sealed envelopes. In long interval misoprostol group, bag (A) contains misoprostol tablets and bag (B) contains placebo tablets. After signing the informed consent, the sequentially numbered sealed envelopes will be opened (according to the sequence of attendance of the patient) by the study nurse. Tablets in bag (A) will be inserted 12 hours before office hysteroscopy and tablets in bag (B) will be inserted 3 hours before office hysteroscopy.
  Interventions: Drug: Long interval misoprostol
- Short interval misoprostol (Active Comparator): A small envelope including two labeled plastic bags (A& B) (each bag containing either 2 misoprostol tablets(400µg) or 2 identically appearing placebo tablets) will be packaged in sequentially numbered sealed envelopes. In short interval misoprostol group, bag (A) contains placebo tablets and bag (B) contains misoprostol tablets. After signing the informed consent, the sequentially numbered sealed envelopes will be opened (according to the sequence of attendance of the patient) by the study nurse. Tablets in bag (A) will be inserted 12 hours before office hysteroscopy and tablets in bag (B) will be inserted 3 hours before office hysteroscopy.
  Interventions: Drug: Short interval misoprostol

INTERVENTIONS:
Drug: Long interval misoprostol — A rigid 2.9 mm hysteroscope with 30° forward oblique lens and outer sheath diameter of 5 mm will be used in the procedure. The uterine cavity will be distended by warm saline at a pressure between 60-80 mmHg. All the procedures will be performed during the proliferative phase using the vaginoscopic approach as described by Betocchi and Selvaggi in 1997. All the procedures will be diagnostic.Pain intensity will be assessed by visual analogue scale during the examination and 30 minutes after the procedure. A visual analogue scale ranging from 0 to 10 will be used (zero indicates no pain and 10 indicates the worst possible experienced pain).
  Other Names: long interval misoprostol group
  Arms: Long interval misoprostol
Drug: Short interval misoprostol — A rigid 2.9 mm hysteroscope with 30° forward oblique lens and outer sheath diameter of 5 mm will be used in the procedure. The uterine cavity will be distended by warm saline at a pressure between 60-80 mmHg. All the procedures will be performed during the proliferative phase using the vaginoscopic approach as described by Betocchi and Selvaggi in 1997. All the procedures will be diagnostic.Pain intensity will be assessed by visual analogue scale during the examination and 30 minutes after the procedure. A visual analogue scale ranging from 0 to 10 will be used (zero indicates no pain and 10 indicates the worst possible experienced pain).
  Other Names: short interval misoprostol group
  Arms: Short interval misoprostol

SUMMARY:
The aim of this study was to determine whether misoprostol administered 12 hours before office hysteroscopy can relieve pain more effectively compared with misoprostol administered 3 hours before office hysteroscopy.

DETAILED DESCRIPTION:
The interval between misoprostol administration and office hysteroscopy may have an influence on its effectiveness in pain reduction. There are limited data on the optimal interval from administration of misoprostol and office hysteroscopy. In previous studies, time interval from administration of misoprostol and office hysteroscopy ranged between 2 hours and 24 hours.

Till now no studies have yet investigated the optimal timing of misoprostol administration prior to office hysteroscopy or operative hysteroscopy. The aim of this study was to determine whether misoprostol administered 12 hours before office hysteroscopy can relieve pain more effectively compared with misoprostol administered 3 hours before office hysteroscopy

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous patients who have an indication for office hysteroscopy

Exclusion Criteria:

* Parous patients, menopausal patients and patients with cervical pathology, and previous cervical surgery will be excluded from the study. Moreover, patients with severe vaginal bleeding, acute pelvic inflammatory disease, glaucoma, allergy to misoprostol, cardiac, liver or kidney diseases

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Intensity of pain | up to 30 minutes

SECONDARY OUTCOMES:
Duration of procedure | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, M.D,PhD, Study Director — Cairo University
Locations (1):
- Obstetrics and Gynecology Department,Cairo university, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Background] Cicinelli E, Rossi AC, Marinaccio M, Matteo M, Saliani N, Tinelli R. Predictive factors for pain experienced at office fluid minihysteroscopy. J Minim Invasive Gynecol. 2007 Jul-Aug;14(4):485-8. doi: 10.1016/j.jmig.2007.03.008. PMID 17630168
- [Derived] Fouda UM, Gad Allah SH, Elshaer HS. Optimal timing of misoprostol administration in nulliparous women undergoing office hysteroscopy: a randomized double-blind placebo-controlled study. Fertil Steril. 2016 Jul;106(1):196-201. doi: 10.1016/j.fertnstert.2016.03.022. Epub 2016 Mar 31. PMID 27037462